CLINICAL TRIAL: NCT02839031
Title: Assessment of a Cognitive-behavioral Group Intervention in Children With Diabetes Mellitus and Their Parents
Brief Title: Cognitive-Behavioral Therapy (CBT) in Children With Diabetes
Acronym: DI-CO
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties (study stopped before the expected 80 inclusions)
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UF 9369
Record Dates: First submitted 2016-07-18; First posted 2016-07-20 (Estimated); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes mellitus; glycaemia; cognitive-behavioral treatment; coping; parents; children
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- "CBT" group (Experimental)
  Interventions: Behavioral: "CBT" (Cognitive-Behavioral Therapy)
- Control group (Sham Comparator)
  Interventions: Behavioral: Control (telephonic support without CBT content)

INTERVENTIONS:
Behavioral: "CBT" (Cognitive-Behavioral Therapy)
  Arms: "CBT" group
Behavioral: Control (telephonic support without CBT content)
  Arms: Control group

SUMMARY:
Diabetes mellitus in children and adolescents is a source of stress and poor quality of life for themselves and their family. Development of adaptive coping strategies may be improved by focused parent and children training. This study assesses a cognitive behavioral treatment (CBT) for children/adolescents with diabetes and their parents in comparison with standard health educational interventions. The investigators main aim is to verify that the CBT program improves overall balance of glycaemia better than phone contact without CBT content (control group). Secondary objectives are expected improvements of health-related quality of life and coping styles in parents and children.

ELIGIBILITY:
Inclusion Criteria:

* Children and teenagers from 6 years-old to 18 years-old
* Having diabetes treated by insulin for at least 1 year
* Followed in pediatric diabetology department of Arnaud de Villeneuve Hospital in University Hospital of Montpellier
* Study Inform Consent signed by both children and parents

Exclusion Criteria:

* Children with developmental delay, severe mental disorders or language delay
* Non French-speaking family
* Children who does not live with at least one of his/her parents
* Children whose residence is not compatible with frequent visits at University Hospital of Montpellier
* Clinical status not compatible with study questionnaires assessment.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 57 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2018-07-01 (Actual)

PRIMARY OUTCOMES:
Glycated hemoglobin (HbA1c) level | up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France